CLINICAL TRIAL: NCT05835180
Title: A Phase I, Open-label, Pharmacokinetic Study of TVB-2640 in Subjects With Mild, Moderate, or Severe Hepatic Impairment Compared to Subjects With Normal Hepatic Function
Brief Title: A Phase I Pharmacokinetic Study of TVB-2640 (Denifanstat) in Subjects With Mild, Moderate, or Severe Hepatic Impairment Compared to Subjects With Normal Hepatic Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sagimet Biosciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SB2640-CLIN-009
Record Dates: First submitted 2023-04-17; First posted 2023-04-28 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Non-alcoholic Steatohepatitis; Hepatic Impairment; Cirrhosis
Keywords: NASH; Hepatic impairment; Cirrhosis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fibrosis | interventions — TVB-2640

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- TVB-2640 50 mg - normal hepatic function (Experimental): Healthy subjects with normal hepatic function receive 50 mg PO daily from Day 1 to Day 4
  Interventions: Drug: TVB-2640 - 50 mg
- TVB-2640 50 mg - mild hepatic function (Experimental): Subjects with mild hepatic impairment will receive 50 mg PO daily from Day 1 to Day 4
  Interventions: Drug: TVB-2640 - 50 mg
- TVB-2640 50 mg - moderate hepatic function (Experimental): Subjects with moderate hepatic impairment will receive 50 mg PO daily from Day 1 to Day 4
  Interventions: Drug: TVB-2640 - 50 mg
- TVB-2640 50 mg - severe hepatic function (Experimental): Subjects with severe hepatic impairment will receive 50 mg PO daily from Day 1 to Day 4
  Interventions: Drug: TVB-2640 - 50 mg

INTERVENTIONS:
Drug: TVB-2640 - 50 mg — TVB-2640 -50 mg administered orally once daily

SUMMARY:
The goal of this phase 1 study is to assess the pharmacokinetics, safety and tolerability following multiple oral doses of TVB-2640 in subjects with mild, moderate, or severe hepatic impairment compared to healthy subjects with normal hepatic function.

ELIGIBILITY:
Key Inclusion Criteria:

Subjects must satisfy all of the following criteria at the Screening visit unless otherwise stated:

All Subjects

* Males or females, of any race, between 18 and 75 years of age, inclusive.
* Body mass index between 18.0 and 42.0/45.0 kg/m2 (inclusive; up to 42.0 kg/m2 for subjects without ascites and 45.0 kg/m2 for subjects with ascites)
* Females will not be pregnant or lactating, and females of childbearing potential (premenopausal females who are anatomically and physiologically capable of becoming pregnant following menarche) and males will agree to use contraception as detailed in the protocol.

Subjects with Hepatic Impairment Only

* Documented chronic stable liver disease; diagnosis of cirrhosis due to parenchymal liver disease. T
* Subjects with mild, moderate, or severe hepatic impairment may have medical findings consistent with their hepatic dysfunction.
* Non-hepatic, abnormal clinical laboratory evaluations must not be clinically relevant.
* Currently on a stable medication regimen; Concomitant medications administered within 30 days prior to the first dose administration (Day 1) must be approved by the Investigator (or designee), Sponsor, and the Medical Monitor.
* Anemia secondary to hepatic disease will be acceptable if hemoglobin > 9 g/dL and anemia symptoms are not clinically significant as judged by the Investigator (or designee) and the Medical Monitor. Subjects must have a platelet count ≥ 35 × 109 platelets/L for mild and moderate hepatic impairment subjects and ≥ 30 × 109 platelets/L for severe hepatic impairment subjects.
* Subjects with diabetes mellitus may be included, provided the subjects have:

  1. Hemoglobin A1c values ≤ 9.0% at Screening. Subjects with values outside this range may be allowed by the Medical Monitor on a case-by-case basis.

Medications for the treatment of diabetes mellitus must be reviewed and approved by the Investigator (or designee), Medical Monitor, and Sponsor.

Key Exclusion Criteria:

Subjects will be excluded from the study if they satisfy any of the following criteria at the Screening visit unless otherwise stated:

All Subjects

* Significant history or clinical manifestation of any metabolic, allergic, dermatological, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the Investigator (or designee).
* History of corneal edema, keratitis, xerophthalmia (dry eye), or other corneal abnormalities. Subjects may wear contact lenses during the study with the exception of the day of dosing (Days 1 to Day 4).
* History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs (except uncomplicated appendectomy, hernia repair, and cholecystectomy will be allowed; bariatric surgery will not be allowed).
* Ventricular dysfunction or history of risk factors for Torsade de Pointes. Subjects will be excluded if there is a family history of long QT syndrome.
* Evidence of hepatorenal syndrome and Cockcroft-Gault estimated creatinine clearance (CrCl) ≤ 60 mL/min/1.73 m2 for mild and moderate hepatic impairment subjects, ≤ 50 mL/min/1.73 m2 for severe hepatic impairment subjects or clinically significant abnormal sodium and potassium levels, as determined by the Investigator (or designee), at Screening or Check-in (Day 1).
* Use or intended use of any medications/products known to alter drug absorption, metabolism, or elimination processes.
* Use of any strong inhibitors or inducers of cytochrome P450 (CYP)2C9 or CYP3A4/5, or inhibitors of CYP3A4 within 30 days prior to first dose administration (Day 1).
* Alcohol consumption of > 21 units per week for males and > 14 units for females.
* Positive urine drug screen
* Positive severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2) polymerase chain reaction (PCR) test at Screening and Check-in (Day -1), history of hospitalization for coronavirus disease-2019 (COVID-19), or history of use of oxygen due to COVID-19. Note that previous COVID-19 infection alone is not exclusionary and vaccination against SARS-CoV-2 is allowed but must be documented.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-12-18 (Actual); Study Completion 2023-12-18 (Actual)

PRIMARY OUTCOMES:
Total TVB-2640 plasma concentration-time (AUC) at steady state | Day 4
  Total TVB-2640 plasma concentration-time curve during a dosing interval at steady-state
Unbound TVB-2640 plasma concentration-time (AUC) at steady state | Day 4
  Unbound TVB-2640 plasma concentration-time curve during a dosing interval at steady-state
Maximum plasma concentration (Cmax) for total TVB-2640 at steady state | Day 4
Maximum plasma concentration (Cmax) for unbound TVB-2640 at steady state | Day 4
incidence and severity of AEs | Screening to Day 7

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - Thomas C. Marbury, Orlando, Florida
  - Eric J. Lawitz, MD, San Antonio, Texas
- Geza Lakner, Kistarcsa, Hungary

IPD SHARING:
Plan to Share IPD: No